CLINICAL TRIAL: NCT01977092
Title: Reducing Offenders' HIV Risk: MI Enhanced Case Management With Drug-Free Housing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health Institute, California (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DA034973-01A1 (NIH); R01DA034973-01A1 (NIH)
Record Dates: First submitted 2013-09-25; First posted 2013-11-06 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-06

CONDITIONS: Alcohol and Drug Abuse
Keywords: sober living houses; HIV; alcohol and drugs
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motivational interviewing case management (Experimental): MICM intervention combines aspects of motivational interviewing along with case management to influence HIV risk and recovery from alcohol and drug problems. Participants assigned to the MICM condition will be contacted to receive 3 individual sessions within the first 4 weeks of entering the study. Thereafter they will have contact with the MICM therapist monthly throughout the duration of their enrollment in the study (12 months).
  Interventions: Behavioral: Motivational interviewing case management
- Resource referrals (Other): Respondents will receive SLH services as usual along with a list of resources that can be used to address a variety of problems.
  Interventions: Behavioral: Resource referrals

INTERVENTIONS:
Behavioral: Motivational interviewing case management
  Arms: Motivational interviewing case management
Behavioral: Resource referrals
  Arms: Resource referrals

SUMMARY:
The goal of the study is to see if a Motivational Interviewing Case Management (MICM) intervention will improve outcomes for respondents who are on probation or parole, at risk for HIV and have recently entered a Sober Living House. The MICM will help respondents access needed services, adapt to their new living environment, find and maintain work, address HIV risk and treatment, and manage setbacks. The risk for HIV infection among criminal justice offenders is significant, as is the need for stable, drug free housing in this population. Our aim is to see if the MICM intervention in the context of drug free housing will improve health outcomes and reduce recidivism.

DETAILED DESCRIPTION:
This study is based on the premise that probationers and parolees must have access to stable, drug-free housing to reduce HIV risk, access needed services and avoid rearrests and reincarceration. Drug-free housing at the Sober Living Network (SLN) in California are being studied as a way to provide a positive living environment for probationers and parolees. The houses use a sober living house (SLH) model of recovery that includes a communal recovery environment, abstinence from drugs and alcohol, peer support, and encouragement to attend self-help groups such as Alcoholics Anonymous.

The proposed study will improve SLHs for offenders by adding a Motivational Interviewing Case Management (MICM) intervention specifically targeted to the problems presented by each offender. The list of potential problems that MICM can address is extensive: 1) adapting to the SLH environment, 2) complying with parole and probation, 3) finding and maintain work, 4) successfully accessing and maintaining retention in services, 5) addressing HIV risk, testing and treatment, 6) mobilizing personal and informal resources, and 7) managing setbacks (e.g., relapse, loss of housing, loss of work).

Men and women involved with the criminal justice system (N=330) entering SLHs will be assigned to a condition consisting of a provision of a resources manual where residents can seek help for a variety of problems (a control group) or the MICM (intervention).To avoid mixing individuals who receive the intervention with individuals who do not within the same house, houses are randomized at the house level. Once a house is randomized to a study condition, all of the individuals recruited from that house receive the same intervention, MICM or SLH as usual. To avoid contamination of study conditions by gender, randomization procedures are stratified by houses for men, women, and both genders. Research interviews are conducted at baseline (within one month of entering the houses), 6 months, and 12 months. Follow-up interviews are conducted whether or not the participant leaves the SLH and at a site that is the most comfortable for the participant.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older
* Speak English
* Entered the sober living house in the last month
* Able to provide contact info for followups
* Willing to attend MICM sessions
* On probation or parole
* ONE of the following: tested positive for HIV, injected drugs, sex work history, men who have sex with men (MSM), or women who have had unprotected sex in the last month with multiple partners

Exclusion Criteria:

* serious mental health disorder that would hinder their ability to provide informed consent or otherwise participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doug Polcin, Ed.D, Principal Investigator — Alcohol Research Group / Public Health Institute
Locations (1):
- Alcohol Research Group, Emeryville, California, United States

REFERENCES:
- See also: Related Info — http://www.arg.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment of 330 study participants followed a two-step process: first we recruited the house, and then we recruited residents that moved in to those houses. The approximately 50 SLHs participating in the study were located in the Los Angeles area and all were members of the Sober Living Network.
Pre-assignment Details: To avoid mixing individuals who received the intervention with individuals who did not within the same house, we randomized at the house level. Once a house was randomized to a study condition, all of the individuals recruited from that house received the same intervention.
Groups:
- Motivational Interviewing Case Management: MICM intervention combines aspects of motivational interviewing along with case management to influence HIV risk and recovery from alcohol and drug problems. Participants assigned to the MICM condition will be contacted to receive 3 individual sessions within the first 4 weeks of entering the study. Thereafter they will have contact with the MICM therapist monthly throughout the duration of their enrollment in the study (12 months).
  Motivational interviewing case management
- Resource Referrals: Respondents will receive SLH services as usual along with a list of resources that can be used to address a variety of problems.
  Resource referrals
Period: Overall Study
Arm/Group | Motivational Interviewing Case Management | Resource Referrals
Started | 149 | 181
Completed | 118 | 151
Not Completed | 31 | 30
Not completed — Death | 3 | 4
Not completed — Lost to Follow-up | 23 | 14
Not completed — Withdrawal by Subject | 2 | 1
Not completed — In prison | 3 | 11

BASELINE CHARACTERISTICS:
Population: Participants in the motivational interviewing case management (MICM) would be set up with their MICM therapist at the end of the baseline interview to set up their first appointment. They would continue with MICM for the 12 months in the study, regardless of whether or not they stayed at the house. The control group was given a list of resources.
Groups:
- Control - Resource Referrals: Respondents will receive sober living house services as usual along with a list of resources that can be used to address a variety of problems.
  control - Resource referrals
- Total: Total of all reporting groups
Arm/Group | Motivational Interviewing Case Management | Control - Resource Referrals | Total
Number analyzed (Participants) | 149 | 181 | 330
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 147 | 179 | 326
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (11.9) | 39.3 (11.6) | 38.1 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 41 | 85
  Male | 105 | 140 | 245
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 44 | 67
  Not Hispanic or Latino | 126 | 137 | 263
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 7
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Black or African American | 46 | 34 | 80
  White | 91 | 126 | 217
  More than one race | 7 | 13 | 20
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 149 | 181 | 330
Legal status [Count of Participants; unit: Participants]
  Probation(including drug court) | 129 | 132 | 261
  Parole | 20 | 49 | 69

OUTCOME MEASURES:

1. Primary Outcome: Change in Criminal Justice Outcomes
Description: Measured by dichotomous measure of whether or not any time spent incarcerated in past 6 months.56 follow-up interviews were conducted in jails, when allowed and the participant was comfortable, but we did not conduct interviews in prison. See participant flow for number of participants in prison.
Time Frame: Baseline, 6 months, and 12 months
Population: 330 participants were interviewed at baseline. We attempted to follow up with all participants, whether or not they stayed at the sober living house, for 6 and 12 month follow up interviews. We were not able to find all of them for follow up interviews.
Measure: Count of Participants; unit: Participants
Groups:
- Control/Resource Referrals: Respondents will receive SLH services as usual along with a list of resources that can be used to address a variety of problems.
  Resource referrals
Arm/Group | Motivational Interviewing Case Management | Control/Resource Referrals
Number analyzed (Participants) | 149 | 181
Participants
  Baseline: Not incarcerated in past 6 months | 66 | 70
  Baseline: Incarcerated in past 6 months | 83 | 111
  6 months: number analyzed (Participants) | 108 | 145
  6 months: Not incarcerated in past 6 months | 94 | 108
  6 months: Incarcerated in past 6 months | 14 | 37
  12 months: number analyzed (Participants) | 118 | 150
  12 months: Not incarcerated in past 6 months | 94 | 105
  12 months: Incarcerated in past 6 months | 24 | 45

2. Primary Outcome: Change in Alcohol and Drug Use (Timeline Follow Back)
Description: Measured by whether or not the participant reports complete abstinence from all substance use for last 6 months on Timeline Followback (TLFB).
Time Frame: Baseline, 6 months, and 12 months
Population: 330 participants were interviewed at baseline. We attempted to follow up with all participants, whether or not they stayed at the sober living house, for 6 and 12 month follow up interviews.
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Interviewing Case Management | Control/Resource Referrals
Number analyzed (Participants) | 149 | 181
Participants
  Baseline: Not abstinent | 100 | 126
  Baseline: Abstinent | 49 | 55
  6 months: number analyzed (Participants) | 108 | 145
  6 months: Not abstinent | 55 | 82
  6 months: Abstinent | 53 | 63
  12 months: number analyzed (Participants) | 118 | 151
  12 months: Not abstinent | 62 | 80
  12 months: Abstinent | 56 | 71

3. Primary Outcome: Change in Worries About HIV in Past 6 Months.
Description: Measured by whether or not the participant was worried about HIV in past 6 months.
Time Frame: Baseline, 6 months, and 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Interviewing Case Management | Control/Resource Referrals
Number analyzed (Participants) | 149 | 181
Participants
  Baseline: Didn't have HIV worry | 25 | 48
  Baseline: Had HIV worry | 124 | 133
  6 months: number analyzed (Participants) | 108 | 145
  6 months: Didn't have HIV worry | 41 | 82
  6 months: Had HIV worry | 67 | 63
  12 months: number analyzed (Participants) | 118 | 151
  12 months: Didn't have HIV worry | 73 | 98
  12 months: Had HIV worry | 45 | 53

ADVERSE EVENTS:
Time Frame: Data was collected for participants for 1 year that they participated in the study.
Description: This study did not involve any medications; participants were randomized to a behavioral intervention. No regular assessments of medical adverse events were collected.This study collected information on Serious Adverse Events in a non-systematic assessment. During the follow up interviews, participants would report the number of hospitalizations in the prior 6 months. The interviewer would then collect additional information for reporting of Serious Adverse Events.
Arm/Group | Motivational Interviewing Case Management | Resource Referrals
All-Cause Mortality (participants affected / at risk) | 3/149 | 4/181
Serious Adverse Events (participants affected / at risk) | 12/149 | 30/181
Other Adverse Events (participants affected / at risk) | 0/149 | 0/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Motivational Interviewing Case Management (N=149) | Resource Referrals (N=181)
Depressive symptoms (Psychiatric disorders) | 1 (1) | 3 (6)
Suicidal symptoms (Psychiatric disorders) | 3 (3) | 15 (27) — Hospitalizations due to suicidal symptoms
Staph infection (General disorders) | 3 (3) | 0 (0)
Contusions and lacerations (General disorders) | 0 (0) | 2 (4)
Cardiac arrhythmia, unspecified (Cardiac disorders) | 0 (0) | 2 (2)
Alcohol withdrawal (General disorders) | 0 (0) | 1 (1)
Unspecified asthma with (acute) exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fracture (General disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 2 (2)
Seizure disorder (Nervous system disorders) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Unconsciousness NOS (General disorders) | 2 (2) | 1 (1)
Gastrointestinal hemorrhage, unspecified (Gastrointestinal disorders) | 0 (0) | 1 (1) — Ppt reported they had internal bleeding due to drug use
Acute embolism and thrombosis of unspecified deep veins of lower extremity (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — ppt reported hospitalization due to a blood clot in leg
Infarction of spleen (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Biliary acute pancreatitis (Endocrine disorders) | 1 (1) | 0 (0)
Contusions (General disorders) | 1 (1) | 0 (0) — Ppt was assaulted and hospitalized overnight due to injuries.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-10-07): https://cdn.clinicaltrials.gov/large-docs/92/NCT01977092/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-07): https://cdn.clinicaltrials.gov/large-docs/92/NCT01977092/SAP_001.pdf